CLINICAL TRIAL: NCT05190315
Title: A Phase I Trial of Chlorpromazine Together With Standard of Care in New Diagnosis of Glioblastoma
Brief Title: Chlorpromazine and Standard of Care in Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mohammed Milhem (Other)
Responsible Party: Sponsor-Investigator, Mohammed Milhem, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202109340
Record Dates: First submitted 2021-12-30; First posted 2022-01-13 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Chlorpromazine; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chlorpromazine with standard of care chemoradiation (Experimental): Each patient will undergo 3 phases of treatment.
  Concurrent Phase: includes concurrent radiation Monday - Friday (60 Gy total radiation dose in 2 Gy fractions), oral temozolomide (75 mg/m2/day) daily for a maximum 49 days starting Day 1 of radiation, and oral chlorpromazine (25 mg for first 3 patients, then escalate to 50 mg if no DLT) daily starting 7 days prior to radiation start.
  Interim Phase: Continue oral chlorpromazine daily dose post-radiation and prior to beginning adjuvant temozolomide.
  Adjuvant Phase: 28 days after radiation fini (+/- 5 business days), Start oral temozolomide (starting dose 150 mg/m2/day and escalated to 200 mg/m2/day if no treatment related adverse events noted) once daily for 5 consecutive days of a 28 day cycle, and continue oral daily chlorpromazine seven days a week per cycle. The adjuvant phase treatment will continue for up to 6 cycles. Cycle length is 28 days.
  Interventions: Drug: Chlorpromazine; Drug: Temozolomide; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Chlorpromazine — Concurrent Phase: Oral chlorpromazine at 25 mg daily for the first 3 patients, then dose escalate to 50 mg if no dose limiting toxicity (DLT). Starting 7 days prior to radiation start.
  Interim Phase: Chlorpromazine, 25 mg per day for first 3 subjects and then dose escalate to 50 mg per day if no DLT, will continue post radiation and prior to beginning adjuvant temozolomide.
  Adjuvant Phase: Chlorpromazine, 25 mg per day for first 3 subjects and then dose escalate to 50 mg per day if no DLT, will be continued daily (7 days per week) concomitant with Temozolomide.
  Other Names: Thorazine
Drug: Temozolomide — Concurrent Phase: Oral temozolomide at 75 mg/m2 per day concomitant with focal radiation and chlorpromazine. Temozolomide should be started on day 1 of radiation therapy, either at bedtime or morning as per patient preference.
  Adjuvant Phase: Oral Temozolomide concomitant with Chlorpromazine, starting Temozolomide dose (Cycle 1) is 150 mg/m2 daily with a single dose escalation to 200 mg/m2 daily in subsequent cycles if no treatment-related adverse events > grade 2 are noted. Temozolomide to be taken once daily for 5 consecutive days (1-5) of a 28 day cycle.
  Other Names: Temodar
Radiation: Radiation Therapy — Concurrent Phase: Radiation therapy administered daily, M-F, to a total dose of 60 Gy in 2 Gy Fractions for a total of 30 fractions.

SUMMARY:
This is a phase 1 study investigating the re-purposing of chlorpromazine, combined with temozolomide and radiation in the treatment of newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
The purpose of the study is to determine the safety and acute toxicity of chlorpromazine (CPZ) when administered throughout the standard treatment protocol for glioblastoma multiforme, as well as determine progression free survival.

Chlorpromazine (25 mg daily for the first 3 patients then dose escalate to 50 mg if no DLT) will be added to a standard of care regimen which includes radiation and adjuvant Temozolomide. Chlorpromazine treatment will continue for up to 6 cycles or until criteria for removal is met. Temozolomide is administered following standard practice adopted at the University of Iowa Hospitals and Clinics (UIHC).

Subject will have several MRI scans for disease assessment throughout the treatment. There will be 3 phases of treatment for each patient:

Concomitant Chlorpromazine- Start 7 days prior to day 1 of concurrent Temozolomide and radiation. Will continue with Chlorpromazine through radiation therapy (temozolomide will cease after 49 days)

Interim Phase- When radiation has ended, subject will take Chlorpromazine for 28 days- no Temozolomide

Adjuvant phase- subject resumes Temozolomide per standard practice, and continues to take Chlorpromazine through 6 cycles of Temozolomide.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed (i.e., within 5 weeks from recent surgery), histologically or cytologically or molecularly confirmed glioblastoma, gliosarcoma, or diffuse midline glioma.
* Diagnosis must be made by surgical biopsy or excision.
* Therapy must begin ≤ 5 weeks after most recent surgery.
* Age ≥ 18 years
* ECOG performance status 0-2 (Karnofsky > 50%, see Appendix B).
* A complete blood count and differential must be obtained within 21 days prior to radiation fraction 1, with adequate bone marrow functions as defined below:

  * Absolute neutrophil count (ANC) ≥ 1500 cells per mm^3
  * Platelets ≥ 100,000 per mm^3
  * Hemoglobin ≥ 8 g/dL
* Plasma blood chemistries within 21 days of radiation fraction 1, as defined below:

  * Creatinine ≤ 2.0 mg/dL
  * Total bilirubin ≤ 1.5 mg/dL
  * ALT ≤ 3 times the institutional upper limit of normal
  * AST ≤ 3 times the institutional upper limit of normal
* Patient or patient's legally authorized representative's ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Recurrent high-grade glioma.
* Significant abnormalities on ECG at screening. QTcF > 450 msec for males or > 470 msec for females at screening.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to temozolomide or chlorpromazine.
* Significant co-morbid central nervous system disease, including but not limited to, multiple sclerosis, Parkinson's disease, history of myasthenia gravis, or dementia.
* Patients with prior malignancies of the same or different tumor type and patients with concurrent malignancies of the same or different tumor type whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational drug.
* Patients who have received prior chemotherapy (including Gliadel wafers) for the current glioma
* Prior radiation therapy to the head or neck, which would result in overlap of radiation therapy fields.
* Patients may not be receiving any other investigational agents. Use of tumor treating fields (TTF) in adjuvant phase is permitted as per standard of care.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, hypoparathyroidism, or psychiatric illness/social situations that would limit compliance with study requirements. Uncontrolled seizures despite being on maximal anti-seizure therapy.
* Pregnant women are excluded from this study because ionizing radiation is a known teratogen, and temozolomide is a Class D agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with temozolomide, breastfeeding should be discontinued if the mother is treated with temozolomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
Safety and acute toxicity of chlorpromazine (CPZ) when administered throughout the standard treatment for glioblastoma multiforme (GBM) will be graded per NCI's Common Terminology Criteria for Adverse Events v 5.0 (CTCAE v5.0) | First treatment through 30 days post last dose of study drug
  The incidence of treatment-emergent adverse events will be summarized by system organ class and/or preferred term, type of adverse event, and severity (based on NCI CTCAE v5.0 grades)
Recommended phase II dose of chlorpromazine in combination with the standard treatment protocol for glioblastoma | 4 weeks
  The study will utilize a 3+3 design, and up to 6 patients will be treated at each dose level. The recommended Phase II dose will be defined as the highest dose level for which at most 1 of 6 patients experience a dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
Progression free survival of patients with newly diagnosed GBM treated with CPZ and standard chemoradiation 6 months from the date of surgery | 2 years
  Time from diagnosis to documented disease progression or death due to any cause.
2-year overall survival of patients with newly diagnosed GBM treated with CPZ and standard chemoradiation 6 months from the date of surgery | 2 years
  Time from diagnosis up to 2 years post completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Milhem, MBBS, Principal Investigator — University of Iowa Hospitals and Clinics Holden Comprehensive Cancer Center
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No